CLINICAL TRIAL: NCT06314867
Title: A Single Center, Randomized, Double-blind, and Intergroup Control Clinical Study to Evaluation on Lot-to-lot Consistency and Immune Persistence of Three Commercial Batches of 23 Valent Pneumococcal Polysaccharide Vaccine
Brief Title: Clinical Study on Lot-to-lot Consistency and Immune Persistence of Three Commercial Batches of PPSV23
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20220231
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-02

CONDITIONS: Healthy Volunteers
Keywords: 23 Valent Pneumococcal Polysaccharide Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 23 Valent Pneumococcal Polysaccharide Vaccine (lot 1) (Experimental): Batch number: Y202112011
  Interventions: Biological: 23 Valent Pneumococcal Polysaccharide Vaccine (lot 1)
- 23 Valent Pneumococcal Polysaccharide Vaccine (lot 2) (Experimental): Batch number: Y202112012
  Interventions: Biological: 23 Valent Pneumococcal Polysaccharide Vaccine (lot 2)
- 23 Valent Pneumococcal Polysaccharide Vaccine (lot 3) (Experimental): Batch number: Y202112013
  Interventions: Biological: 23 Valent Pneumococcal Polysaccharide Vaccine (lot 3)

INTERVENTIONS:
Biological: 23 Valent Pneumococcal Polysaccharide Vaccine (lot 1) — All subjects were vaccinated with 1 dose of 23 Valent Pneumococcal Polysaccharide Vaccine (batch number: Y202112011), intramuscularly injected into the lateral deltoid muscle of the upper arm.
  Arms: 23 Valent Pneumococcal Polysaccharide Vaccine (lot 1)
Biological: 23 Valent Pneumococcal Polysaccharide Vaccine (lot 2) — All subjects were vaccinated with 1 dose of 23 Valent Pneumococcal Polysaccharide Vaccine (batch number: Y202112012), intramuscularly injected into the lateral deltoid muscle of the upper arm.
  Arms: 23 Valent Pneumococcal Polysaccharide Vaccine (lot 2)
Biological: 23 Valent Pneumococcal Polysaccharide Vaccine (lot 3) — All subjects were vaccinated with 1 dose of 23 Valent Pneumococcal Polysaccharide Vaccine (batch number: Y202112013), intramuscularly injected into the lateral deltoid muscle of the upper arm.
  Arms: 23 Valent Pneumococcal Polysaccharide Vaccine (lot 3)

SUMMARY:
The research objective is to evaluate lot-to-lot consistency and immune persistence of three commercial batches of 23 valent pneumococcal polysaccharide vaccine.

DETAILED DESCRIPTION:
This study adopted a randomized, double-blind, equivalency design with different batches of experimental vaccine. 990 individuals aged 18-59 were included and divided into three groups at a ratio of 1:1:1, with 330 individuals in each group receiving three batches of experimental vaccines, respectively. All subjects were vaccinated with 1 dose of 0.5ml, intramuscularly injected into the lateral deltoid muscle of the upper arm.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 18-59;
* Voluntarily participate and sign an informed consent form;
* Subjects are able to comply with the requirements of the clinical study protocol and complete the prescribed follow-up;
* Has not received pneumococcal vaccine or any other preventive products recently (has not received attenuated live vaccine within 14 days, has not received inactivated vaccine within 7 days);
* Underarm temperature ≤ 37.0 ℃;
* Female participants of childbearing age agree to take effective contraceptive measures within 3 months from the start of the study until the full vaccination period.

Exclusion Criteria:

* Subjects with a history or family history of progressive neurological disorders such as epilepsy, encephalopathy, and mental illness;
* Has a history of severe allergies to any drugs or vaccines in the past;
* Has a allergy history to any component of the experimental vaccine (the main components of the vaccine include type 23 pneumococcal polysaccharides, sodium chloride, sodium dihydrogen phosphate, and sodium dihydrogen phosphate);
* Suffering from severe cardiovascular diseases (heart disease, pulmonary heart disease, pulmonary edema, drug-resistant hypertension (systolic blood pressure ≥ 160mmHg and/or diastolic blood pressure ≥ 100mmHg)); drug-resistant diabetes;
* Subjects with a history of thrombocytopenia or other coagulation disorders that may cause contraindications for subcutaneous injection;
* Subjects with known immunological dysfunction or low levels, or HIV infection;
* Any situation leading to splenomegaly, splenectomy, or functional splenomegaly;
* Malignant tumors, active or treated tumors that have not been clearly cured, or are likely to recur during the study period;
* Anti tuberculosis prevention or treatment is under way;
* Subjects who are participating in or planning to participate in clinical trials of other drugs or vaccine clinical trials throughout the entire observation period;
* Women of childbearing age are in pregnancy (positive urine pregnancy test) or lactation period;
* Any situation that the researcher believes may affect the evaluation of the study.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 990 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Geometric mean concentration (GMC) levels | 30 days after immunization
  Geometric mean concentration (GMC) levels of 23 serotype specific IgG antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Lin Du, Study Chair — Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd
Locations (1):
- Sichuan Center for Disease Control and Prevention, Chengdu, Sichuan, China